CLINICAL TRIAL: NCT04798950
Title: Bronchi Dilation in Polynesian Patients: Monocentric Retrospective Study
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Centre Hospitalier Intercommunal Creteil (Other)
Responsible Party: Sponsor
Other Study IDs: POLYDEB
Record Dates: First submitted 2021-03-11; First posted 2021-03-16 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Polynesian Bronchiectasis
Keywords: bronchi dilatation
MeSH Terms: conditions — Kartagener Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study hypothesis is that dilations of idiopathic bronchi are particularly common in French Polynesia, and that there are arguments in favour of an underlying genetic factor.

The study will retrieve retrospective data in the history of bronchial dilation, patients' personal and family history, microbiological and scannographic data, and the latest cardio respiratory checkup.

ELIGIBILITY:
Inclusion Criteria:

* Polynesian patient
* Patient with bronchial dilation followed by Centre hospitalier de Polynesie Francaise or patient with bonchial dilation no longer consulting in the hospital over the study period Jan 1, 2010 to Dec 31, 2020

Exclusion Criteria:

* Expressed refusal to participate in the study for patients undergoing follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 500 patients with bronchial dilatation over the study period: Jan 1, 2010 to Dec 31, 2020
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2023-06-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Describe the detailed phenotype of bronchi dilation in the Polynesian population | Day 1
  * Clinical criteria: age of onset, personal or family history, smoking Changes in respiratory function
  * Infectious complications: types of bronchial colonization (bacterial, mycobacterial and mycological)
  * Scantographic aspect: Appearance of bronchectasis: cylindrical, varicose orcious, cystic Distributions: LSD, LM, LID, LSG, LIG

SECONDARY OUTCOMES:
Highlighting indirect arguments for a genetic cause | Day 1
  Age of onset of symptoms, frequency of so-called "idiopathic" bronchi dilatation, frequency of inbreeding, familial history